CLINICAL TRIAL: NCT06171048
Title: A Pharmacokinetics Study of CM310 Recombinant Humanized Monoclonal Antibody Injection in Healthy Subjects
Brief Title: Study Evaluating the Pharmacokinetics of CM310 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM310-100005
Record Dates: First submitted 2023-12-05; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): CM310 injection, Subcutaneous
  Interventions: Biological: CM310
- Group B (Experimental): CM310 injection, Subcutaneous
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — CM310 injection

SUMMARY:
This is a single-center, randomized, open-label study to evaluate the pharmacokinetics of CM310 in healthy subjects.

DETAILED DESCRIPTION:
This study includes screening and treatment and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* 20 years ≤ age ≤ 45 years.
* Voluntarily participate in the study and sign the ICF.
* Have the ability to understand the study.

Exclusion Criteria:

* With history of chronic or serious illness.
* With any medication within 28 days prior to administration;
* Plan to undergo surgery during the research period;
* With any situations unsuitable to participate in this study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic: the maximum concentration (Cmax) | up to week 6
  Concentration and exposure

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China